CLINICAL TRIAL: NCT01543412
Title: Folfiri as Second-Line Chemotherapy for Advanced Pancreatic Cancer. A GISCAD Phase II Study
Brief Title: Second Line Chemotherapy for Advanced Pancreatic Cancer
Acronym: SLAP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Italiano per lo studio dei Carcinomi dell'Apparato Digerente (Other)
Collaborators: Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-004637-16
Record Dates: First submitted 2010-09-07; First posted 2012-03-05 (Estimated); Last update posted 2012-03-05 (Estimated); Status verified 2012-02

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: FOLFIRI; Metastases; pancreatic adenocarcinoma; locally advanced or metastatic pancreatic adenocarcinoma
MeSH Terms: conditions — Neoplasm Metastasis | interventions — IFL protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FOLFIRI (Experimental): Folfiri consist of Irinotecan 180 mg/m2 iv on day 1, Leucovorin(l-form) 200 mg/m2 iv on day 1and 2, 5-FU 400 mg/m2 iv bolus on day 1and 2, 5-FU 600 mg/m2 iv by ci for 22 hours on day 1 and 2, repeated every 2 wks The use of antiemetic prophylaxis was decided locally.
  Interventions: Drug: FOLFIRI

INTERVENTIONS:
Drug: FOLFIRI — Irinotecan 180 mg/m2 iv on day 1, Leucovorin(l-form) 200 mg/m2 iv on day 1,2 5-FU 400 mg/m2 iv bolus on day 1,2 5-FU 600 mg/m2 iv by ci for 22 hrs on day 1,2 repeated every 2 wks

SUMMARY:
No validated second-line chemotherapy for the treatment of locally advanced/metastatic pancreatic cancer is actually available,after the failure of a gemcitabine(+/- Cisplatin or Oxaliplatin)-based regimen.

Irinotecan seems to be a moderately active drug in the treatment of this disease Recently was reported some interesting results using a potentially non -cross resistant regimen (FOLFIRI) which could be useful even as second-line chemotherapy.

An exploratory study in this setting seem warranted.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent prior to beginning protocol specific procedures
* Previous chemotherapy with Gemcitabine plus or less Platinoids
* Previous gemcitabine delivered as a radiosensitizer for locally advanced disease, followed or not by a gemcitabine plus or less platinoids as maintenance or disease progression is allowed.
* Male or female less than 75 years of age
* Diagnosis of histologically or cytologically confirmed adenocarcinoma of the pancreas
* Locally advanced (non-resectable) or metastatic pancreatic cancer
* Presence of at least one uni-dimensional indicator lesion measurable by CT scan or MRI in not an irradiated area
* ECOG performance status 0 to 1 at study entry
* Life expectancy: more than 3 months
* Neutrophils more than 1.5 x 109L, platelets more than 100 x 109L, and hemoglobin more than 10 gdL
* Bilirubin level either normal or less than 1.5 x ULN
* ASAT and ALAT normal or less than 2.5 x ULN (normal or less than 5 x ULN if liver metastasis are present)
* Serum creatinine less than 1.5 x ULN
* Amylase normal or less than 1.5 ULN
* Effective contraception for both male and female patients if the risk of conception exists
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be assessed with the patient before registration in the trial

Exclusion Criteria:

* Brain metastases
* Previous treatment with irinotecan or fluoropyrimidines
* Significant cardiovascular disease: clinically relevant coronary artery disease or a history of a myocardial infarction within the last 6 months
* Significant gastrointestinal abnormalities
* Gilbert's Syndrome
* Any uncontrolled infections
* Known HIV infection
* Radiotherapy within 4 weeks prior to study entry
* Any investigational agents 4 weeks prior to entry
* Known grade 3 or 4 allergic reaction to any of the components of the treatment
* Known drug abuse or alcohol abuse
* Medical or psychological condition which in the opinion of the investigator would not permit the patient to complete the study or sign meaningful informed consent
* Women who are pregnant or breastfeeding
* Any concurrent malignancy other than non-melanoma skin cancer, or carcinoma in situ of the cervix.
* Legal incapacity or limited legal capacity

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-01; Primary Completion 2011-06 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (RECIST Criteria) | 2 years
  time from randomization date to date of death from any cause

SECONDARY OUTCOMES:
Safety and tolerability; Safety (CTC criteria - version 3.0) | 18 months
  Treatment will consist of 4 combination-chemotherapy cycles and in case of stable or responsive disease, other 4 cycles can be administered at investigator's discretion. Therefore will be administered for up to 6 months Each treatment cycle will consist of 2 weeks, unless the start of the subsequent cycle is delayed, in which case the cycle length will be longer than 4 weeks.
Overall survival (OS) | time from first cycle to death
  OS is calculated using the Kaplan-Meyer method The principal objective of the trial is to assess the therapeutic activity of FOLFIRI in patients with exocrine pancreas carcinoma.
  The primary activity parameter to be determined is overall response rate.
Progression Free Survival | time from first cycle to progression or death
  PFS was calculated using the Kaplan-Meyer method Presence of at least one target lesion measurable by CT scan or MRI in not an irradiated area (and conform with the RECIST criteria)

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Zaniboni, MD, Study Chair — Fondazione GISCAD; Roberto Labianca, MD, Principal Investigator — Fondazione GISCAD
Locations (9):
- Italy (9):
  - Ospedali Riuniti Umberto I - GM Lancisi-G Salesi, Ancona, Ancona
  - Ospedali Riuniti, Largo Barozzi, 1, Bergamo, Bergamo
  - A.O. Treviglio-Caravaggio, P.le Ospedale n1, Treviglio, Bergamo
  - Fondazione Poliambulanza, Via Bissolati 57, Brescia, Brescia
  - Azienda Ospedaliera "Di Liegro", Gaeta, Latina
  - A.O. Carlo Poma - Via Albertoni, 1, Mantova, Mantova
  - A.O. Ospedale S.Paolo, Milan, MI
  - A.O. S.Salvatore, Pesaro, PS
  - Ospedale Morelli, Sondalo, SO

REFERENCES:
- [Derived] Zaniboni A, Aitini E, Barni S, Ferrari D, Cascinu S, Catalano V, Valmadre G, Ferrara D, Veltri E, Codignola C, Labianca R. FOLFIRI as second-line chemotherapy for advanced pancreatic cancer: a GISCAD multicenter phase II study. Cancer Chemother Pharmacol. 2012 Jun;69(6):1641-5. doi: 10.1007/s00280-012-1875-1. Epub 2012 May 11. PMID 22576338